CLINICAL TRIAL: NCT03955484
Title: The Relationship of Lower Urinary System Symptoms Due to Benign Prostatic Hyperplasia and Urinary Glycosaminoglycan Level
Brief Title: Benign Prostatic Hyperplasia and Glycosaminoglycan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Cagri Akin Sekerci, Urologist, Principal Investigator, MD, Marmara University
Other Study IDs: MAR.UAD.005
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Prostatic Hyperplasia
Keywords: Prostatic Hyperplasia; Lower Urinary Tract Symptoms; Medical Treatment; Urine Marker; Glycosaminoglycan
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who had benign prostatic hyperplasia: Male patients presenting with lower urinary tract symptoms to urology outpatient clinic
  According to the European Association of Urology Guidelines:
  International prostate symptom score> 8 Prostate volume> 40 ml Q max <15 ml /sn Patients who did not receive any treatment for lower urinary tract symptoms and applied for the first time Patients who have not undergone lower urinary tract surgery
  Interventions: Diagnostic Test: Urinary Glycosaminoglycan

INTERVENTIONS:
Diagnostic Test: Urinary Glycosaminoglycan — Urine will be collected from patients before and after one month of medical treatment (alpha-blocker). After being centrifuged at 5000 g for 10 minutes, urine will be stored at -80 ° C. At the end of the study, urinary glycosaminoglycan levels will be studied by spectrophotometric method.

SUMMARY:
Lower urinary tract symptoms (LUTS) are one of the most common conditions in the urology clinic, affecting at least one in four men after 40 years of age. Benign prostatic hyperplasia is the most common cause of LUTS. Bladder dysfunction (hypersensitivity or detrusor overactivity) and bladder outlet obstruction are two main pathologies involved in the etiology of LUTS. In men aged 40-49, moderate and severe LUTS are reported as 26%, while this ratio is doubled in the age group of 70 years and older. Clinically, BPH is defined as an international symptom score of more than 8, a prostate volume of more than 30 ml, and a maximum flow rate of less than 15 ml / sec. Alpha blockers are recommended as the first-line medical treatment according to European Urology Guidelines (EAU Guidelines 2018) for patients diagnosed with BPH clinically. In recent years, many studies have been published on the relationship of urinary biomarkers with LUTS. Nerve growth factor and brain derived neurotrophic factor have been shown to be closely related to neurogenic or non-neurogenic detrusor overactivity and significant improvements were observed after treatment.The relationship between urinary glycosaminoglycan and overactive bladder has been shown and it has been reported that the values have decreased after treatment.Male patients with LUTS caused by BPH often have symptoms of overactive bladder. However, as far as we know, there is no study in the literature about the meaning of urinary GAG levels in this patient group. The aim of this study was to investigate the relationship between urinary glycosaminoglycan levels and patients who had benign prostatic hyperplasia with and without overactive bladder symptoms.

DETAILED DESCRIPTION:
35 patients and 10 controls were planned to be included in the study. Urine will be collected from patients before and after one month of medical treatment (alpha-blocker). After being centrifuged at 5000 g for 10 minutes, urine will be stored at -80 ° C. At the end of the study, urinary glycosaminoglycan levels will be studied by spectrophotometric method. Urine GAG levels and pre and post treatment uroflowmetry, IPSS, overactive bladder symptom score, bladder frequency volume chart, post void residual urine volume will be compared.

ELIGIBILITY:
Eligibility Criteria

1. Male patients presenting with lower urinary tract symptoms to urology outpatient clinic
2. According to the European Association of Urology Guidelines:

   1. International prostate symptom score> 8
   2. Prostate volume> 40 ml
   3. Q max <15 ml /sn
3. Patients who did not receive any treatment for lower urinary tract symptoms and applied for the first time
4. Patients who have not undergone lower urinary tract surgery

Exclusion Criteria

1. Patients who had undergone medical and surgical treatment for lower urinary tract symptoms
2. Patients with accompanying urethral stricture
3. Patients with neurological diseases (Parkinson's, Multiple Sclerosis etc ...)
4. Patients with spinal cord trauma
5. Patients with indication for surgical treatment at the time of initial admission (Macroscopic hematuria, bladder stone, urinary retention, upper urinary tract dilatation)

Ages: 40 Years to 70 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients who had benign prostatic hyperplasia with and without overactive bladder symptoms.
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
The value of glycosaminoglycan in predicting the success of medical treatment of benign prostatic hyperplasia | one month

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang LW, Han XM, Chen CH, Ma Y, Hai B. Urinary brain-derived neurotrophic factor: a potential biomarker for objective diagnosis of overactive bladder. Int Urol Nephrol. 2014 Feb;46(2):341-7. doi: 10.1007/s11255-013-0540-x. Epub 2013 Aug 28. PMID 23982767
- [Background] Bhide AA, Cartwright R, Khullar V, Digesu GA. Biomarkers in overactive bladder. Int Urogynecol J. 2013 Jul;24(7):1065-72. doi: 10.1007/s00192-012-2027-1. Epub 2013 Jan 12. PMID 23314226
- [Background] Suh YS, Ko KJ, Kim TH, Lee HS, Sung HH, Cho WJ, Lee KS. Urinary Nerve Growth Factor as a Potential Biomarker of Treatment Outcomes in Overactive Bladder Patients. Int Neurourol J. 2017 Dec;21(4):270-281. doi: 10.5213/inj.1732794.397. Epub 2017 Dec 31. PMID 29298466
- [Background] Alkis O, Zumrutbas AE, Toktas C, Aybek H, Aybek Z. The use of biomarkers in the diagnosis and treatment of overactive bladder: Can we predict the patients who will be resistant to treatment? Neurourol Urodyn. 2017 Feb;36(2):390-393. doi: 10.1002/nau.22939. Epub 2015 Dec 10. PMID 26661444
- [Background] Mashima R, Sakai E, Tanaka M, Kosuga M, Okuyama T. The levels of urinary glycosaminoglycans of patients with attenuated and severe type of mucopolysaccharidosis II determined by liquid chromatography-tandem mass spectrometry. Mol Genet Metab Rep. 2016 Apr 22;7:87-91. doi: 10.1016/j.ymgmr.2016.03.009. eCollection 2016 Jun. PMID 27331006
- [Background] Siracusano S, Cucchi A, Ciciliato S, Lampropoulou N, Vittur F. Urinary levels of glycosaminoglycans in patients with idiopathic detrusor overactivity. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Dec;20(12):1477-80. doi: 10.1007/s00192-009-0973-z. Epub 2009 Aug 12. PMID 19672549